CLINICAL TRIAL: NCT01201330
Title: Retrospective Cohort Study of ONJ
Brief Title: DPBRN Retrospective Cohort Study of Osteonecrosis of the Jaw
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: HealthPartners Institute (Other); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Gregg H. Gilbert, DDS, MBA, Study Chair, University of Alabama at Birmingham
Other Study IDs: 106030; U01DE016747 (NIH)
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Osteonecrosis of the Jaw
Keywords: ONJ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ONJ sufferers: history of jaw osteonecrosis
- Bisphosphonate exposure: patients with exposure to bisphosphonates

SUMMARY:
The purpose of this study was to determine the prevalence of ONJ in the patient population of 2 large HMOs and study the risk factors associated with the development of this condition.

DETAILED DESCRIPTION:
The electronic database from Kaiser Permanente and HealthParnters of Minnesota were used to identify all ONJ cases that occured between 1994 and 2006 and then demographic, social and medical risk factors possibly associated with the disease were abstracted and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* ONJ sufferers and control biphosphonate users older than 40, of any gender, race and ethnic origin

Min Age: 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients older than 40 with a history of jaw osteonecrosis and control patients with exposure to biphosphonates were included.
Sampling Method: Non-Probability Sample
Enrollment: 572606 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Fellows, Ph.D., Principal Investigator — Kaiser Permanente; Andrei Barasch, DMD,MDSc, Principal Investigator — University of Alabama at Birmingham; Brad Rindal, DMD, Principal Investigator — HealthPartners of Minnesota; Gregg H Gilbert, DDS, MBA, Study Chair — University of Alabama School of Dentistry
Locations (1):
- Gregg H. Gilbert, DDS, MBA, Birmingham, Alabama, United States